CLINICAL TRIAL: NCT04028453
Title: Follow up of Increased Nuchal Translucency :Study of 2010 to 2018 of Limoges Hospital
Acronym: HYPERCLAIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI19_0030 (HYPERCLAIR)
Record Dates: First submitted 2019-07-15; First posted 2019-07-22 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Ultrasound Fetal Medicine
Keywords: Increased nuchal translucency; prenatal diagnosis; karyotype analysis; chromosome micro-array analysis; neurodevelopmental disorders; euploid children
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mother: There will be a first part with a retrospective study in order to collect pregnancy data to answer to the primary endpoint. Then, there will be a prospective part where mothers and their children will have to answer an evaluation questionnaire.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — There will be a first part with a retrospective study in order to collect pregnancy data to answer to the primary endpoint. Then, there will be a prospective part where mothers and their children will have to answer an evaluation survey.

SUMMARY:
The ultrasound of the first trimester allows to determinate the pregnancy beginning, the type of pregnancy and also to detect increased nuchal translucency (NT). Fetuses with common chromosomal abnormalities (trisomies 21, 18 and 13 and monosomy X) and structural abnormalities (particularly cardiac defects) and single-gene disorders frequently show increased NT. The purpose of this study is to evaluate in the population of Limousin, the type and frequency of these abnormalities.

DETAILED DESCRIPTION:
Increased NT superior than 95th percentile (Nicolaides curves) during the ultrasound of the first trimester, are associated to common chromosomal abnormalities. It's therefore necessary to make amniocentesis and to analyze karyotyping and Genomic microarrays, also known as chromosomal microarrays (CMA). In euploid foetus, increased NT is also associated with structural defects or genetic syndromes. Additionally, the overall long-term growth of euploid children with increased NT is not much known. The majority (98%) of euploid children with a normal second trimester ultrasound is apparently healthy in the short run. The investigator's objective is to evaluate in a retrospective way, different events (structural defects, chromosomal or genetic abnormalities) during these pregnancies. In a prospective way, the neurodevelopmental disorders in euploid children will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Increased nucal translucency (NT) > 95e percentile on the pregnancy's first trimester
* Monofoetal pregnancy
* Twin pregnancy (biamniotic bichorial)
* Adult patients

Exclusion Criteria:

* Increased NT < 95e percentile on the pregnancy's first trimester
* Increased NT > 95e percentile on the pregnancy's second trimester
* Twin pregnancy (biamniotic monochorial), triple or more gestation
* Underage patients

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patient with nuchal translucency of the fetus> 95th percentile in the first trimester of pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Number of chromosomal abnormalities on fetuses with increased nuchal translucency | 6 months
  Characterization of fetuses with increased nuchal translucency by Identification of chromosomal abnormalities, structural defects and genetic syndromes on fetuses with increased nuchal translucency
Number structural defects on fetuses with increased nuchal translucency | 6 months
  Characterization of fetuses with increased nuchal translucency by Identification of chromosomal abnormalities, structural defects and genetic syndromes on fetuses with increased nuchal translucency
Number of genetic syndromes on fetuses with increased nuchal translucency | 6 months
  Characterization of fetuses with increased nuchal translucency by Identification of chromosomal abnormalities, structural defects and genetic syndromes on fetuses with increased nuchal translucency

SECONDARY OUTCOMES:
Rate of each Pregnancy outcomes | 1 year
  Numbers of alive children, fetal death in utero, abortions on medical grounds, stillborn, children born prematurely
structural defects | 1 year
  Numbers and type term of structural defects
maternofetal infection | 1 year
  number and type of maternofetal infection
postnatal structural defects | 1 year
  Numbers and type of postnatal structural defects
postnatal chromosomal abnormalities | 1 year
  Number and type of postnatal chromosomal abnormalities
postnatal genetic syndromes | 1 year
  Number and type of postnatal genetic syndromes
Determination of a neck thickness threshold at risk of psychomotor developmental delay | 1 year
  Neurodevelopmental evaluation score of Age Stage Questionnaire ASQ-3 (for 2 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years children) or Global School Adaptation GSA (from 6 to 8 years children).
Determination of a neck thickness threshold at risk of malformations and requiring the persistence of monthly ultrasound monitoring | 1 year
  Numbers and type of postnatal structural defects
Study of the psychomotor development of nuchal translucency with normal genetic analysis | 1 year
  Neurodevelopmental evaluation score of Age Stage Questionnaire (ASQ-3) (for 2 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years children without genetic abnormalities) or Global School Adaptation (GSA) (from 6 to 8 years children without genetic abnormalities).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No